CLINICAL TRIAL: NCT06029010
Title: Real-world Study in Metastatic Colorectal Cancer Patients With Long-term Responses to Regorafenib in the US
Brief Title: An Observational Study to Learn More About the Long-Term Responses to Treatment With Regorafenib in Patients With Metastatic Colorectal Cancer in the United States
Acronym: COLONGER
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22624
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Colorectal Cancer
Keywords: mCRC
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Long-term responders of regorafenib ≥5 months: Defined as treatment duration ≥5 months after treatment initiation.
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506)
- Long-term responders of regorafenib ≥4 months: Defined as treatment duration ≥4 months after treatment initiation.
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506)

INTERVENTIONS:
Drug: Regorafenib (Stivarga, BAY73-4506) — Follow clinical administration.

SUMMARY:
This is an observational study in which data already collected from patients with metastatic colorectal cancer will be studied.

Metastatic colorectal cancer (mCRC) is a cancer of the colon (large bowel) or the rectum (lowest part of the bowel just before the anus) that has spread to other parts of the body.

The study drug, regorafenib, is already approved for cancer doctors to prescribe to patients with mCRC. It is an anti-cancer drug that blocks several proteins, called enzymes, which are involved in the growth of cancer.

The participants in this study were treated with regorafenib as part of their regular care from their doctors.

Some studies have shown that patients with mCRC who took regorafenib had improved survival outcomes, and some of them did well on the treatment for a long time. Cancer doctors have also reported from their routine practice that some patients with mCRC are able to respond to regorafenib for a longer period than others. However, there is limited knowledge about which people this is likely to happen for.

To better understand the long-term response of regorafenib treatment, there is a need for a large-scale study in the real world.

The main purpose of this study is to learn more about patients who showed a long-term response to regorafenib as a mono treatment for mCRC. To do this, researchers will collect the following information from the participants' health records:

Duration of treatment with regorafenib

Percentage of participants who received treatment with regorafenib for at least 5 months and 4 months.

Characteristics, including age, sex, race, health condition, and signs and symptoms of mCRC, of participants who received treatment with regorafenib for at least 5 months and 4 months.

The data will come from an electronic health records database called the Flatiron Health Data Repository for patients in the United States. The data will be from patients with mCRC who started treatment with regorafenib between July 2013 and December 2022.

Researchers will consider the data of the participants collected until May 2023.

In this study, only available data from routine care are collected. No visits or tests are required as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of mCRC between 1 JAN 2013 and 31 DEC 2022 who initiated regorafenib monotherapy up to 14 days prior or after mCRC diagnosis and during the patient selection period (1 JUL 2013 to 31 DEC 2022).
* Adult patients (≥18 years old) at index date (date of first regorafenib treatment).
* Patients with at least one recorded visit, laboratory test, or other recorded electronic medical record (EMR) entry (e.g., treatment) in the Flatiron network at least 3 months prior to the index date, unless the patient was diagnosed with mCRC within the last 3 months.

Exclusion Criteria:

* Patients who had a diagnosis or recorded history of gastrointestinal stromal tumor (GISC), hepatocellular cancer (HCC), or other primary cancers (except non-melanoma skin cancers) during the 6-month period on or prior to the index date.
* For analyses of long-term responders, patients will be excluded if treatment duration <5 and <4 months for treatment completers, or treatment duration <5 and <4 months at last visit date for non-completers.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data for the study will be obtained from the Flatiron Health Data Repository; an electronic health record (EHR)-derived longitudinal demographically and geographically diverse database of oncology patients in routine clinical practice in the US.
  Patients with mCRC who initiated regorafenib treatment between 1 JUL 2013 and 31 DEC 2022 will be followed through the electronic data from the start of regorafenib treatment until the date of death for patients who died, and the date of last visit on or up to 31 MAY 2023 for patients with no record of death.
Sampling Method: Non-Probability Sample
Enrollment: 2326 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
Duration of treatment with regorafenib monotherapy in patients who had a long-term response to regorafenib monotherapy, as indicated by a treatment duration of ≥5 months | Retrospective analysis from 01-Jan-2013 to 31-May-2023
Demographic characteristics of patients who had a long-term response to regorafenib monotherapy, as indicated by a treatment duration of ≥5 months | Retrospective analysis from 01-Jan-2013 to 31-May-2023
Descriptive analysis of clinical characteristics of patients who had a long-term response to regorafenib monotherapy, as indicated by a treatment duration of ≥5 months | Retrospective analysis from 01-Jan-2013 to 31-May-2023
Descriptive analysis of biomarkers of patients with mCRC who had a long-term response to regorafenib monotherapy, as indicated by a treatment duration of ≥5 months | Retrospective analysis from 01-Jan-2013 to 31-May-2023

SECONDARY OUTCOMES:
Duration of treatment with regorafenib monotherapy in patients who had a long-term response to regorafenib monotherapy, as indicated by a treatment duration of ≥4 months | Retrospective analysis from 01-Jan-2013 to 31-May-2023
Demographic characteristics of patients who had a long-term response to regorafenib monotherapy, as indicated by a treatment duration of ≥4 months | Retrospective analysis from 01-Jan-2013 to 31-May-2023
Descriptive analysis of clinical characteristics of patients who had a long-term response to regorafenib monotherapy, as indicated by a treatment duration of ≥4 months | Retrospective analysis from 01-Jan-2013 to 31-May-2023
Descriptive analysis of biomarkers of patients with mCRC who had a long-term response to regorafenib monotherapy, as indicated by a treatment duration of ≥4 months | Retrospective analysis from 01-Jan-2013 to 31-May-2023

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.